CLINICAL TRIAL: NCT00904358
Title: Validity and Reliability of Non-invasive Estimation of Central Venous Pressure by Measurement of Internal Jugular Size Using 2-dimensional Ultrasound
Brief Title: Estimation of Internal Jugular Vein Central Venous Pressure (CVP) by Ultrasound
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: Si183/2009
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Internal Jugular Size Measured by Ultrasound; Central Venous Pressure
Keywords: internal jugular vein; cross sectional area; ultrasound; central venous pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- cross sectional area: internal jugular cross sectional area measured by ultrasound
  Interventions: Diagnostic Test: cross sectional area

INTERVENTIONS:
Diagnostic Test: cross sectional area

SUMMARY:
To study the validity and reliability of estimation of the central venous pressure by measurement of internal jugular vein size using 2-dimensional ultrasound.

DETAILED DESCRIPTION:
Objectives:

1. To study the validity and reliability of estimation of the central venous pressure by measurement of internal jugular vein size using 2-dimensional ultrasound.
2. To evaluate the correlation of internal jugular vein cross sectional area and central venous pressure.

Methods:

1. The study design is prospective observational study.
2. We will include all patients scheduled for cardiac surgery in Siriraj Hospital and record both internal jugular size using 2-dimensional ultrasound just before central venous catheter insertion. The central venous pressure will be recorded and the ultrasound picture will be measured.
3. The data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for cardiac surgery
* need central venous catheterization intraoperatively
* elective surgery
* age > 18

Exclusion Criteria:

* neck pathology
* history of internal jugular or SVC thrombosis
* limited neck mobility
* severe valvular lesion
* decompensated heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for cardiac surgery in Siriraj Hospital
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
internal jugular size | 1 day
  Cross-sectional area of internal jugular vein measured by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Kasana Raksamani, MD, Principal Investigator — Mahidol University
Locations (2):
- Thailand (2):
  - Faculty of Medicine, Siriraj Hospital, Bangkok
  - Kasana Raksamani, Bangkok